CLINICAL TRIAL: NCT06481228
Title: Efficacy and Safety of Molecular Targeted Therapy Combined With Chemotherapy and Sequential CAR-T Cells in Newly Diagnosed Adult Patients With Philadelphia Chromosome-Positive B-cell Acute Lymphoblastic Leukemia
Brief Title: Efficacy and Safety of TKI Combined With Chemotherapy and Sequential CAR-T Cells in ND Adult Patients With Ph+ ALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024019
Record Dates: First submitted 2024-05-24; First posted 2024-07-01 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Philadelphia Positive Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia, Adult
Keywords: Ph-Positive Acute Lymphoblastic Leukemia; CAR-T cell; Venetoclax; olverembatinib; Newly Diagnosed
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Immunotherapy, Adoptive; venetoclax; olverembatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TKI Combined With Chemotherapy and Sequential CAR-T Cells (Experimental): Ph+ALL patients receiving CAR-T cells as consolidation therapy after achieving complete remission (CR) with overembatinib, venetoclax and reduced-intensity chemotherapy.
  Interventions: Combination Product: CAR-T cells; Drug: Venetoclax; Drug: Olverembatinib

INTERVENTIONS:
Combination Product: CAR-T cells — CAR-T cells as consolidation therapy
Drug: Venetoclax — BCL2 inhibitor
Drug: Olverembatinib — TKI

SUMMARY:
In recent years, immunotherapy (eg. blinatumomab, inotuzumab ozogamicin, CAR-T cells) has demonstrated a high safety and efficacy profile in relapsed/refractory (R/R）B-ALL. The available data suggest that the advancement of immunotherapy from R/R field to the frontline setting may be an important approach to increase the depth of remission, which ultimately translates into a survival benefit. In this study, the investigators propose a treatment regimen using CAR-T cell therapy as a consolidation method for Ph+ ALL patients achieving complete remission (CR) with overembatinib, venetoclax and reduced-intensity chemotherapy, aiming to reduce the total cycles of chemotherapy and related toxicities, shorten length of hospitalization, and ultimately improve patients' survival and quality of life.

DETAILED DESCRIPTION:
The CAR-T cells were murine-derived second-generation CD19 CAR-T with a co-stimulation domain of 4-1BB, and the infusion dose was 1×10^6/kg CAR+ cells in a single infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or older
2. Newly diagnosed Philadelphia chromosome positive(either t(9;22) and/or BCR-ABL positive and/ or FISH positive) acute lymphoblastic leukemia
3. CD19 expression on blasts
4. Expected survival time greater than 3 months
5. Adequate end organ function as defined by: Total bilirubin ≤ 1.5 x upper limit of normal（ULN）; serum alanine aminotransferase (ALT) and serum aspartate aminotransferase (AST) ≤ 2.5 x ULN or ≤5 x ULN if leukemic involvement of the liver is present; Creatinine ≤ 1.5 x ULN; Serum amylase and lipase ≤ 1.5 x ULN; Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related; normal electrolytes: Potassium ≥ LLN; Magnesium ≥ LLN; Phosphorus ≥ LLN; Cardiac color Doppler ultrasound ejection fraction ≥ 45%
6. Subject has provided written informed consent prior to any screening procedure

Exclusion Criteria:

1. Lymphoid blast crisis of chronic myelocytic leukemia (CML)
2. Previous or ongoing systemic anti-ALL therapy (including but not restricted to TKI and/or radiotherapy, except for appropriate pre-treatment)
3. Patients with a history of myocardial infarction within 12 months or clinically significant cardiac disorders disease (e.g., unstable angina, congestive heart failure, uncontrollable hypertension, uncontrollable arrhythmia, etc.)
4. Uncontrolled active serious infections that could, in the investigator's opinion, potentially interfere with the completion of treatment
5. Known HIV seropositivity
6. History of acute pancreatitis within 1 year of study screening or history of chronic pancreatitis
7. Uncontrolled hypertriglyceridemia (triglycerides >450 mg/dL)
8. Another malignancy diagnosed and treated within 5 years prior to diagnosis or previously diagnosed with another malignancy with evidence of residual disease. Patients with non-melanoma skin cancer or any type of carcinoma in situ that has been completely excised should not be excluded
9. Female patients who are pregnant or breast feeding
10. Clinical manifestations of active CNS or extramedullary involvement with ALL
11. Poorly controlled diabetes, defined as glycosylated hemoglobin (HbA1c) values of >7.5%. Patients with preexisting, well-controlled diabetes are not excluded
12. Any serious psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment
13. Other conditions assessed by the investigators to be inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) | Up to 2 years post-registration
  From CR1 to relapse, death from any cause or last follow-up

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years post-registration
  From the date of registration to the date of death resulting from any cause.
Event-free survival (EFS) | Up to 5 years post-registration
  From the date of registration to the date of induction failure, relapse, death from any cause, or last follow-up
Cumulative rate of complete molecular response | Up to 1 year post-registration
  The cumulative rate of patients achieving complete molecular remission
MRD-negative complete remission rate measured by NGS tracking clonal IG/TR rearrangements | Up to 1 year post-registration
  No clonal IG/TR rearrangements were detected by NGS
Cumulative incidence of relapse (CIR) | Up to 2 years post-registration
  Calculated with the cumulative incidence method, with death in patients who had a complete hematologic response as a competing risk.
The rate of adverse | Up to 5 years post-registration
  adverse events during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China